CLINICAL TRIAL: NCT01481246
Title: The Neurocognitive Study for the Aging
Brief Title: Neurocognitive Study for the Aging-a Longitudinal Study With a Greek Cypriot Cohort
Acronym: NEUROAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Fofi Constantinidou, Professor, University of Cyprus
Other Study IDs: Humanities/Society/0308(ΒΕ)/07; Humanities/Society/0308(ΒΕ)/07 (Other Grant/Funding Number: Cyprus Research Promotion Foundation); SKEPSH (Other Grant/Funding Number: European Regional Development Fund); EXCELLENCE/1216/0404 (Other Grant/Funding Number: Cyprus Research Innovation Foundation)
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Aging; Memory Impairment; Cognitive Decline; Mild Cognitive Disorder
Keywords: neurorehabilitation; cognition; aging; MCI; cognitive decline
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — APOE phenotyping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal Aging/Cognitive Decline: Health adults as well as adults with MCI and early stage AD are being recruited in the study
  Interventions: Behavioral: Categorization training; Behavioral: Psychosocial and Psychoeducational Group training

INTERVENTIONS:
Behavioral: Categorization training — Behavioral intervention consisting of cognitive training exercises to improve categorization performance
Behavioral: Psychosocial and Psychoeducational Group training — Group treatment with a focus on psychosocial and psychoeducational intervention in healthy adults and in adults with cognitive decline. Ten week cycle, 2 hours per week group intervention study.

SUMMARY:
The Neurocognitive Study for the Aging (NEUROAGE) was initially funded by the Cyprus Innovation Foundation and has received subsequent funding by the European Union Regional Development Fund. The project focuses on the understanding of the effects of age on neurocognitive abilities such as attention, memory, language, categorization, and executive functioning. In addition, specific arms of the project investigate the effects of a theory-driven hierarchical training program, the Categorization Program, to improve cognitive abilities in adults with Mild Cognitive Impairment (MCI) and of a group intervention program focusing on cognitive and psychosocial abilities. Over 1000 adults ages 40 and older have been recruited in the NEUROAGE project thus far. The grant was awarded to the University of Cyprus, with Professor Fofi Constantinidou as the PI.

DETAILED DESCRIPTION:
Given the fact that older adults are expected to live longer while maintaining their social and professional activities, the development of effective cognitive retraining methodologies designed to maximize independence has been of interest. In addition to changes caused by the normal aging process, older adults over 65 are at a high risk for developing dementia. About 8-12% of the older adult population will demonstrate a pre-dementia syndrome referred to as Mild Cognitive Impairment (MCI) which is considered a prodrome to dementia. Consequently, it is important to identify variables that contribute to the development of MCI as well as neurocognitive therapy approaches to help patients improve their level of functioning.

Categorization is one of the most fundamental cognitive processes. The ability to divide the world into discrete categories is a rudimentary process beginning early in life and continues to be developed and refined across the lifespan. This underlying process is crucial to a variety of neurocognitive abilities including attention and memory and can influence vocational and educational reintegration. Normal aging results in categorization deficits which in turn can interfere with the individual's ability to attend, remember, and organize information. This difficulty could hamper activities of daily living, social participation, and independence. This project implements an innovative treatment program based on current theoretical models of human cognition designed to improve neurocognitive abilities.

One of the objectives of the project is to provide evidence on the effectiveness of a systematic and hierarchical neurocognitive therapy method, the Categorization Program (CP) in adults with MCI and in normal older adults. It is hypothesized that the CP will be an effective treatment approach to improve categorization abilities in both groups of subjects. In addition, since 2020, we have been implementing a group intervention program as part of our recent funding to investigate its feasibility in healthy older adults and in adults with MCI.

The following activities have been taking place:

1. Initially, a population-based sample of 500 older adults was tested using a battery of neuropsychological measures. Normal older adults are reassessed every two years. Currently, more than 800 healthy adults have been recruited in this project.
2. Second, normal OA and adults with MCI have been randomly assigned into either the treated or untreated groups. The treated groups receive the CP training in order to test its effectiveness.
3. Third, the long term effects of cognitive retraining is being assessed.
4. Finally, the project examines the relationship between the categorization tasks, neuropsychological performance, functional outcome measures, and subject characteristics including health indices, education, and biomarkers. Theoretical constructs such as Cognitive Reserve have been explored as part of this project.

The long-term objective of this research program is to determine variables that influence cognitive decline in older adults and develop effective neurocognitive therapy techniques.

ELIGIBILITY:
Inclusion Criteria:

* healthy with no prior neurological history

Exclusion Criteria:

* prior neurological history or significant psychiatric history

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal older adults and adults with cognitive decline are recruited in this study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Tests | on going
  a variety of cognitive tests as well as psychosocial measures are used in this project

CONTACTS AND LOCATIONS:
Overall Officials: Fofi Constantinidou, Ph.D., Principal Investigator — University of Cyprus
Locations (1):
- University of Cyprus, Nicosia, Cyprus

REFERENCES:
- [Derived] Chadjikyprianou A, Constantinidou F. Effectiveness of a Novel Multidimensional Group Intervention to Enhance Subjective Cognitive and Psychosocial Functioning in Healthy Older Adults. J Aging Health. 2025 Oct 24:8982643251391224. doi: 10.1177/08982643251391224. Online ahead of print. PMID 41135181
- [Derived] Chadjikyprianou A, Constantinidou F. A new multidimensional group intervention for cognitive and psychosocial functioning for older adults: Background, content, and process evaluation. Front Med (Lausanne). 2023 Apr 20;10:1161060. doi: 10.3389/fmed.2023.1161060. eCollection 2023. PMID 37153102
- See also: Center for Applied Neuroscience — http://www.cancyprus.org